CLINICAL TRIAL: NCT02040402
Title: Comparison of the Immunogenicity of the 3+1 Schedule and the 2+1 Schedule of 7-valent Pneumococcal Conjugated Vaccine in Young Chinese Infants
Brief Title: Immunogenicity of 3+1 Versus 2+1 Schedule for PCV7
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Society for the Relief of Disabled Children, Hong Kong (Unknown)
Responsible Party: Principal Investigator, Lau Yu Lung, Chair Professor of Paediatrics, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 09-024
Record Dates: First submitted 2013-12-19; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Infectious Disease
Keywords: Comparison of pneumococcal conjugated vaccine regimes
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4-Dose Regimen (Active Comparator): 3+1 schedule of 7-valent pneumococcal conjugated vaccine:
  Infants who are randomized for 3+1 schedule will be administrated one dose of PCV7 at the age of 2 months old, 4months old and 6 months old. A booster dose will be administrated at the age of 12 months old.
  Infants will be followed up for 12-16 months starting from vaccination of first dose. There is no restriction on the use of other medications before or during the follow-up period.
  Interventions: Biological: 7-valent pneumococcal conjugated vaccine
- 3-Dose Regimen (Active Comparator): 2+1 schedule of 7-valent pneumococcal conjugated vaccine:
  Infants who are randomized for 2+1 schedule will be administrated with one dose of PCV7 at the age of 2 months old and 4months old. A booster dose will be administrated at the age of 12 months old.
  Infants will be followed up for 12-16 months starting from vaccination of first dose. There is no restriction on the use of other medications before or during the follow-up period.
  Interventions: Biological: 7-valent pneumococcal conjugated vaccine

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugated vaccine — Pneumococcal vaccine 3+1 and 2+1 schedule comparison
  Arms: 3-Dose Regimen
Biological: 7-valent pneumococcal conjugated vaccine — 3+1 doses vs 2+1 doses
  Arms: 4-Dose Regimen

SUMMARY:
Pneumonia is one of the most prevalent diseases in infants and children. The incidence of pneumonia in children less than 5 years old is about 34-40 cases per 1000 in Europe and America and more than 2 million children die of pneumonia annually. It was reported that Streptococcus pneumoniae accounted for 13%-53% of lower respiratory tract infections in different age group of infants or children. In addition, 7%-9% of bacterial meningitis was due to Streptococcus pneumoniae infection. In addition, children infected with Streptococcus pneumoniae often transmit the pathogens to adult. As a result, it is evident that Streptococcus pneumoniae presents a heavy burden to paediatrics practice.

Vaccination of 7-valent pneumococcal conjugate vaccines is effective in preventing Streptococcus pneumonia .Routine use of PCV7 in the US has rapidly reduced rates of invasive pneumococcal disease in children. The impact of the vaccine was noted within 1 year of introduction. According to Centre for Disease Control's (CDC) Active Bacterial Core Surveillance (ABCs) the incidence of invasive pneumococcal disease among children <5 years dropped 75% from 1998/1999 to 2005; disease caused by vaccine-type strains fell 94% from 80 to 4.6 per 100,000. Currently there are two immunization schedules: manufacturer recommended the 3+1 schedule and many countries adopted a 3 dose schedule, either 3+0 or 2+1 schedules. In US, it is recommended to give three doses during infancy (scheduled at 2, 4, 6 month) plus one dose at 12-15 months (3+1 schedule). Since several studies have demonstrated that two doses may provide similar direct protection to three conjugate doses during infancy, it is recommended to give two doses during infancy plus a booster dose 12 months in some European countries including United Kingdom.

In this trial, the immunogenicity of the 3+1 schedule and the 2+1 schedule of 7-valent pneumococcal conjugated vaccine in young infants will be compared.

DETAILED DESCRIPTION:
Streptococcus pneumonia is the most common bacterial pathogen of community-acquired pneumonia in children [1]. It may also cause meningitis, bloodstream infections and acute otitis media [1]. In 2005, WHO estimated that 1.6 million people a year die from pneumococcal disease, including up to 1 million children less than 5 years old worldwide, in particularly for infants and children less than 2 years old [1]. Most of the death occur in developing countries [2, 3]. Case fatality ratios are highest for invasive infections and range from 5-20% for bacteremia to 40-50% for meningitis. Among meningitis survivors, long-term neurologic sequelae occur in 25-56% of cases [4].

Most pneumococcal infections can be treated effectively with antibiotics, although meningitis still often results in devastating outcomes. Over the last 20 years, the emergence of antimicrobial resistance among S. pneumoniae complicates treatment of infections. Penicillin and co-trimoxazole resistance are common in many parts of the world, including China [5-9]. Multidrug resistance has also emerged and is best documented in industrialized countries. Treatment failures due to resistance have been documented for acute otitis media, meningitis and bloodstream infections [5-6].

Currently two pneumococcal vaccines are licensed and available. One is the 23-valent pneumococcal polysaccharide vaccine (PPV23). However it is not recommended for children less than 2 year old. Another one is the 7-valent pneumococcal conjugate vaccine (PCV7) which can be used for children 6 weeks to 24 months of age. PCV7 includes the capsular polysaccharide of 7 serotypes (4,6B, 9V, 14, 18C, 19F, 23F), each coupled to a nontoxic variant of diphtheria toxin, CRM197. The vaccine contains 2 μg each of capsular polysaccharide from serotypes 4,9V, 14, 19F and 23F; 2 μg of oligosaccharide from 18C; 4 μg of capsular polysaccharide of 6B; 20 μg of CRM197; and 0.125 mg of aluminum/0.5 ml dose as an aluminum phosphate adjuvant [10].

Since the licensure of the PCV7 in 2000, it is being widely used for infants and toddlers in most of the developed countries. It has been demonstrated that PCV7 provide great protections for pneumococcal invasive disease (meningitis, bloodstream infections), pneumonia and otitis media [11, 12]. Routine use of PCV7 in the US has rapidly reduced rates of invasive pneumococcal disease in children. The impact of the vaccine was noted within 1 year of introduction. According to CDC's Active Bacterial Core Surveillance (ABCs) the incidence of invasive pneumococcal disease among children <5 years dropped 75% from 1998/1999 to 2005; disease caused by vaccine-type strains fell 94% from 80 to 4.6 per 100,000 [13, 14]. A multi-centre study of hospitalized patients found that 77% fewer cases in children <2 years were caused by vaccine serotypes in 2002 compared to the average number of cases during 1994-2000 [15]. Surveillance data on vaccine impact from outside the US are currently limited. Data from Calgary, Canada showed a 93% reduction in vaccine-type invasive disease in children <2 years of age [16]. In Australia, the rate of vaccine-type invasive pneumococcal disease reduced by 78% between 2002 and 2006 in children aged under 2 years [17]. In US, it was also found that one or more doses of PCV7 was 96% effective against invasive disease in healthy children, 81% effective in children with comorbid medical conditions and 76% effective overall against disease caused by strains resistant to penicillin [18]. PCV7 use also appears to be reducing non-invasive pneumococcal infections in the US, including otitis media and pneumonia [19-22].

Currently there are two immunization schedules: the 3+1 and the 2+1 schedules. In US, it is recommended to give three doses during infancy (scheduled at 2, 4, 6 month) plus one dose at 12-15 months (3+1 schedule). Since several studies have demonstrated that two doses may provide similar direct protection to three conjugate doses during infancy, it is recommended to give two doses during infancy plus a booster dose 12 months in some European countries including UK [23, 24].

In China, a recent serogroup distribution study in out-patient department (OPD) patients with acute upper respiratory infections showed that coverage with PCV7 was about 55% for nasopharyngeal carriage pneumococci isolates, and 75% for the penicillin-nonsusceptible pneumococci isolates from 2000 to 2005 [25], suggesting that PCV7 is effective for preventing pneumococcal infections. Since PCV7 was only licensed in China by May of 2008, there is no data for the effectiveness. For immunization schedule, the manufacturer of PCV7 (Wyeth Pharmaceuticals Inc) recommends to use 3+1 schedule in China as that in US. However, China may NOT have enough resources for mass vaccination as a developing country because PCV7 is very expensive. Therefore, generating our own data in China and developing an alternative immunization schedule, such as 2+1, may have great advantage to save more lives by using a limited resource.

ELIGIBILITY:
Inclusion Criteria:

Chinese infants born in Hong Kong

Exclusion Criteria:

(i)Previous administration of PCV7 or other pneumococcal vaccines

(ii)History of immunodeficiency

(iii)Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment

(iv)Malignancy, other than squamous cell or basal cell skin cancer

(v)Autoimmune disease

(vi)History of asthma or reactive airways disease

(vii)Cardiovascular and pulmonary disorder, chronic metabolic disease (including diabetes), renal dysfunction or hemoglobinopathies requiring regular medical follow-up or hospitalization during the preceding year

(viii)Use of immunosuppressive medication

(ix)Receipt of blood products or immunoglobulin in the past 6 month

Ages: 6 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Serological response in terms of geometric mean titres after the primary dose series and booster for the 2+1 and 3+1 schedules. | An average of one month post vaccination

SECONDARY OUTCOMES:
Proportion of infants with Immunoglobulin G concentrations above 0.35ug/ml to the 7 serotypes | An average of one month post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yu-lung LAU, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Pneumococcal conjugate vaccine for childhood immunization--WHO position paper. Wkly Epidemiol Rec. 2007 Mar 23;82(12):93-104. No abstract available. English, French. PMID 17380597
- [Background] Black RE, Morris SS, Bryce J. Where and why are 10 million children dying every year? Lancet. 2003 Jun 28;361(9376):2226-34. doi: 10.1016/S0140-6736(03)13779-8. PMID 12842379
- [Background] Bryce J, Boschi-Pinto C, Shibuya K, Black RE; WHO Child Health Epidemiology Reference Group. WHO estimates of the causes of death in children. Lancet. 2005 Mar 26-Apr 1;365(9465):1147-52. doi: 10.1016/S0140-6736(05)71877-8. PMID 15794969
- [Background] Goetghebuer T, West TE, Wermenbol V, Cadbury AL, Milligan P, Lloyd-Evans N, Adegbola RA, Mulholland EK, Greenwood BM, Weber MW. Outcome of meningitis caused by Streptococcus pneumoniae and Haemophilus influenzae type b in children in The Gambia. Trop Med Int Health. 2000 Mar;5(3):207-13. doi: 10.1046/j.1365-3156.2000.00535.x. PMID 10747284
- [Background] Mera RM, Miller LA, Daniels JJ, Weil JG, White AR. Increasing prevalence of multidrug-resistant Streptococcus pneumoniae in the United States over a 10-year period: Alexander Project. Diagn Microbiol Infect Dis. 2005 Mar;51(3):195-200. doi: 10.1016/j.diagmicrobio.2004.10.009. PMID 15766606
- [Background] Whitney CG, Farley MM, Hadler J, Harrison LH, Lexau C, Reingold A, Lefkowitz L, Cieslak PR, Cetron M, Zell ER, Jorgensen JH, Schuchat A; Active Bacterial Core Surveillance Program of the Emerging Infections Program Network. Increasing prevalence of multidrug-resistant Streptococcus pneumoniae in the United States. N Engl J Med. 2000 Dec 28;343(26):1917-24. doi: 10.1056/NEJM200012283432603. PMID 11136262
- [Background] Kyaw MH, Lynfield R, Schaffner W, Craig AS, Hadler J, Reingold A, Thomas AR, Harrison LH, Bennett NM, Farley MM, Facklam RR, Jorgensen JH, Besser J, Zell ER, Schuchat A, Whitney CG; Active Bacterial Core Surveillance of the Emerging Infections Program Network. Effect of introduction of the pneumococcal conjugate vaccine on drug-resistant Streptococcus pneumoniae. N Engl J Med. 2006 Apr 6;354(14):1455-63. doi: 10.1056/NEJMoa051642. PMID 16598044
- [Background] Song JH, Lee NY, Ichiyama S, Yoshida R, Hirakata Y, Fu W, Chongthaleong A, Aswapokee N, Chiu CH, Lalitha MK, Thomas K, Perera J, Yee TT, Jamal F, Warsa UC, Vinh BX, Jacobs MR, Appelbaum PC, Pai CH. Spread of drug-resistant Streptococcus pneumoniae in Asian countries: Asian Network for Surveillance of Resistant Pathogens (ANSORP) Study. Clin Infect Dis. 1999 Jun;28(6):1206-11. doi: 10.1086/514783. PMID 10451154
- [Background] Yao K, Shen X, Yul S, Lu Q, Deng L, Ye Q, Zhang H, Deng Q, Hu Y, Yang Y. Antimicrobial resistance and serotypes of nasopharyngeal strains of Streptococcus pneumoniae in Chinese children with acute respiratory infections. J Int Med Res. 2007 Mar-Apr;35(2):253-67. doi: 10.1177/147323000703500210. PMID 17542413
- [Background] Murray D, Jackson C. A conjugate vaccine for the prevention of pediatric pneumococcal disease. Mil Med. 2002 Aug;167(8):671-7. PMID 12188240
- [Background] Trotter CL, McVernon J, Ramsay ME, Whitney CG, Mulholland EK, Goldblatt D, Hombach J, Kieny MP; SAGE subgroup. Optimising the use of conjugate vaccines to prevent disease caused by Haemophilus influenzae type b, Neisseria meningitidis and Streptococcus pneumoniae. Vaccine. 2008 Aug 18;26(35):4434-45. doi: 10.1016/j.vaccine.2008.05.073. Epub 2008 Jun 17. PMID 18617296
- [Background] Trotter CL, Greenwood BM. Meningococcal carriage in the African meningitis belt. Lancet Infect Dis. 2007 Dec;7(12):797-803. doi: 10.1016/S1473-3099(07)70288-8. PMID 18045562
- [Background] Whitney CG, Farley MM, Hadler J, Harrison LH, Bennett NM, Lynfield R, Reingold A, Cieslak PR, Pilishvili T, Jackson D, Facklam RR, Jorgensen JH, Schuchat A; Active Bacterial Core Surveillance of the Emerging Infections Program Network. Decline in invasive pneumococcal disease after the introduction of protein-polysaccharide conjugate vaccine. N Engl J Med. 2003 May 1;348(18):1737-46. doi: 10.1056/NEJMoa022823. PMID 12724479
- [Background] Centers for Disease Control and Prevention (CDC). Direct and indirect effects of routine vaccination of children with 7-valent pneumococcal conjugate vaccine on incidence of invasive pneumococcal disease--United States, 1998-2003. MMWR Morb Mortal Wkly Rep. 2005 Sep 16;54(36):893-7. PMID 16163262
- [Background] Kaplan SL, Mason EO Jr, Wald ER, Schutze GE, Bradley JS, Tan TQ, Hoffman JA, Givner LB, Yogev R, Barson WJ. Decrease of invasive pneumococcal infections in children among 8 children's hospitals in the United States after the introduction of the 7-valent pneumococcal conjugate vaccine. Pediatrics. 2004 Mar;113(3 Pt 1):443-9. doi: 10.1542/peds.113.3.443. PMID 14993532
- [Background] Kellner JD, Church DL, MacDonald J, Tyrrell GJ, Scheifele D. Progress in the prevention of pneumococcal infection. CMAJ. 2005 Nov 8;173(10):1149-51. doi: 10.1503/cmaj.051150. No abstract available. PMID 16275962
- [Background] Roche PW, Krause V, Cook H, Barralet J, Coleman D, Sweeny A, Fielding J, Giele C, Gilmour R, Holland R, Kampen R; Enhanced Invasive Pneumococcal Disease Surveillance Working Group; Brown M, Gilbert L, Hogg G, Murphy D; Pneumococcal Working Party of the Communicable Diseases Network Australia. Invasive pneumococcal disease in Australia, 2006. Commun Dis Intell Q Rep. 2008 Mar;32(1):18-30. doi: 10.33321/cdi.2008.32.3. PMID 18522302
- [Background] Mahon BE, Hsu K, Karumuri S, Kaplan SL, Mason EO Jr, Pelton SI; U.S. Pediatric Multicenter Pneumococcal Surveillance Group; Massachusetts Department of Public Health Epidemiologists. Effectiveness of abbreviated and delayed 7-valent pneumococcal conjugate vaccine dosing regimens. Vaccine. 2006 Mar 24;24(14):2514-20. doi: 10.1016/j.vaccine.2005.12.025. Epub 2005 Dec 27. PMID 16417951
- [Background] Whitney CG, Pilishvili T, Farley MM, Schaffner W, Craig AS, Lynfield R, Nyquist AC, Gershman KA, Vazquez M, Bennett NM, Reingold A, Thomas A, Glode MP, Zell ER, Jorgensen JH, Beall B, Schuchat A. Effectiveness of seven-valent pneumococcal conjugate vaccine against invasive pneumococcal disease: a matched case-control study. Lancet. 2006 Oct 28;368(9546):1495-502. doi: 10.1016/S0140-6736(06)69637-2. PMID 17071283
- [Background] Poehling KA, Szilagyi PG, Grijalva CG, Martin SW, LaFleur B, Mitchel E, Barth RD, Nuorti JP, Griffin MR. Reduction of frequent otitis media and pressure-equalizing tube insertions in children after introduction of pneumococcal conjugate vaccine. Pediatrics. 2007 Apr;119(4):707-15. doi: 10.1542/peds.2006-2138. PMID 17403841
- [Background] Grijalva CG, Poehling KA, Nuorti JP, Zhu Y, Martin SW, Edwards KM, Griffin MR. National impact of universal childhood immunization with pneumococcal conjugate vaccine on outpatient medical care visits in the United States. Pediatrics. 2006 Sep;118(3):865-73. doi: 10.1542/peds.2006-0492. PMID 16950975
- [Background] Grijalva CG, Nuorti JP, Arbogast PG, Martin SW, Edwards KM, Griffin MR. Decline in pneumonia admissions after routine childhood immunisation with pneumococcal conjugate vaccine in the USA: a time-series analysis. Lancet. 2007 Apr 7;369(9568):1179-86. doi: 10.1016/S0140-6736(07)60564-9. PMID 17416262
- [Background] Esposito S, Lizioli A, Lastrico A, Begliatti E, Rognoni A, Tagliabue C, Cesati L, Carreri V, Principi N. Impact on respiratory tract infections of heptavalent pneumococcal conjugate vaccine administered at 3, 5 and 11 months of age. Respir Res. 2007 Feb 21;8(1):12. doi: 10.1186/1465-9921-8-12. PMID 17313667
- [Background] Goldblatt D, Southern J, Ashton L, Richmond P, Burbidge P, Tasevska J, Crowley-Luke A, Andrews N, Morris R, Borrow R, Cartwright K, Miller E. Immunogenicity and boosting after a reduced number of doses of a pneumococcal conjugate vaccine in infants and toddlers. Pediatr Infect Dis J. 2006 Apr;25(4):312-9. doi: 10.1097/01.inf.0000207483.60267.e7. PMID 16567982
- [Background] Yu S, Yao K, Shen X, Zhang W, Liu X, Yang Y. Serogroup distribution and antimicrobial resistance of nasopharyngeal isolates of Streptococcus pneumoniae among Beijing children with upper respiratory infections (2000-2005). Eur J Clin Microbiol Infect Dis. 2008 Aug;27(8):649-55. doi: 10.1007/s10096-008-0481-y. Epub 2008 Mar 18. PMID 18347822